CLINICAL TRIAL: NCT04450134
Title: Role of Histamine H1/H2 Receptors in the Health- and Performance-promoting Adaptations to High-intensity Interval Training
Brief Title: Histamine H1/H2 Receptors and Training Adaptations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HIST-TRAINING (BC-06009)
Record Dates: First submitted 2020-06-09; First posted 2020-06-29 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Exercise Training; Physical Activity
Keywords: Exercise; Physiology
MeSH Terms: conditions — Motor Activity | interventions — Lactose; fexofenadine; Famotidine; High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Placebo + exercise vs histamine blockade + exercise
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind for researchers and participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 6 weeks high-intensity interval training + placebo intake
  Interventions: Other: Lactose; Other: High-intensity interval training (HIIT)
- Blockade (Experimental): 6 weeks high-intensity interval training + histamine H1/H2 receptor blockade
  Interventions: Drug: Fexofenadine Hydrochloride; Drug: Famotidine; Other: High-intensity interval training (HIIT)

INTERVENTIONS:
Other: Lactose — Placebo: Lactose capsules
  Arms: Placebo
Drug: Fexofenadine Hydrochloride — H1 receptor antagonist: 540 mg Fexofenadine Hydrochloride
  Arms: Blockade
Drug: Famotidine — H2 receptor antagonist: 40 mg Famotidine
  Arms: Blockade
Other: High-intensity interval training (HIIT) — 6 weeks HIIT

SUMMARY:
Exercise training is beneficial for both health and performance. Histamine has been shown to be involved in the acute exercise response. The current study addresses the role of histamine H1/H2 receptor signaling in the chronic training-induced adaptations. Results from this study will yield more insights into the molecular mechanisms of adaptations to exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary or low levels of physical activity
* Caucasian

Exclusion Criteria:

* Chronic diseases
* Medication use
* Smoking
* Excessive alcohol consumption
* Seasonal allergies

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness | Before, after 3 weeks and after 6 weeks of exercise training
  Change in maximal oxygen uptake during incremental cycling test on cycle ergometer during the 6 week training period
Change in peak aerobic power output | Before, after 3 weeks and after 6 weeks of exercise training
  Change in peak power output during incremental cycling test on cycle ergometer during the 6 week training period
Change in whole-body insulin sensitivity | Before and after 6 weeks of exercise training
  Change from baseline in Matsuda index for whole-body insulin sensitivity derived from Oral Glucose Tolerance Test after the 6 week training period
Change in microvascular function | Before and after 6 weeks of exercise training
  Change from baseline in microvascular function (Single Passive Leg Movement technique) after the 6 week training period

SECONDARY OUTCOMES:
Change in skeletal muscle capillarization | Before and after 6 weeks of exercise training
  Change from baseline in skeletal muscle capillarization (immunohistochemistry) after the 6 week training period
Change in skeletal muscle enzyme activity | Before and after 6 weeks of exercise training
  Change from baseline in enzyme activity assessment of markers of relevance for skeletal muscle function after the 6 week training period
Change in skeletal muscle protein content | Before and after 6 weeks of exercise training
  Change from baseline in Western Blot assessment of markers of relevance for skeletal muscle function after the 6 week training period
Change in power output at Gas Exchange Threshold (GET) | Before, after 3 weeks and after 6 weeks of exercise training
  Change from baseline in GET during incremental cycling test after the 6 week training period
Change in power output at Respiratory Compensation Point (RCP) | Before, after 3 weeks and after 6 weeks of exercise training
  Change from baseline in RCP during incremental cycling test after the 6 week training period
Change in time to exhaustion performance test | Before, after 3 weeks and after 6 weeks of exercise training
  Change in time to exhaustion test (performed after incremental cycling test) during the 6 week training period
Change in heart rate during submaximal cycling | Before and after 6 weeks of exercise training
  Change from baseline in heart rate during submaximal cycling after the 6 week training period
Change in substrate oxidation during submaximal cycling | Before and after 6 weeks of exercise training
  Change from baseline in substrate oxidation during submaximal cycling test (estimated via gas exchange data) after the 6 week training period
Change in blood lactate accumulation during submaximal cycling | Before and after 6 weeks of exercise training
  Change from baseline in capillary lactate concentration at end of submaximal cycling test after the 6 week training period
Change in cycling efficiency during submaximal cycling | Before and after 6 weeks of exercise training
  Change from baseline in cycling efficiency (estimated via gas exchange data) after the 6 week training period
Change in fasted serum insulin concentrations | Before and after 6 weeks of exercise training
  Change from baseline in fasted blood concentrations of insulin after the 6 week training period
Change in fasted serum glucose concentrations | Before and after 6 weeks of exercise training
  Change from baseline in fasted blood concentrations of glucose after the 6 week training period
Change in fasted serum cholesterol concentrations | Before and after 6 weeks of exercise training
  Change from baseline in fasted blood concentrations of cholesterol after the 6 week training period
Change in fasted serum triglyceride concentrations | Before and after 6 weeks of exercise training
  Change from baseline in fasted blood concentrations of triglyceride after the 6 week training period
Change in resting blood pressure | Before and after 6 weeks of exercise training
  Change from baseline in resting mean arterial blood pressure after the 6 week training period
Change in resting heart rate | Before and after 6 weeks of exercise training
  Change from baseline in resting heart rate after the 6 week training period
Change in body weight | Before and after 6 weeks of exercise training
  Change from baseline in total body weight after the 6 week training period

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Movement and Sports Sciences, Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided